CLINICAL TRIAL: NCT07259200
Title: Assessment of Sleep Parameters Using Polygraphy in Patients With Paroxysmal Atrial Fibrillation Qualified for Pulmonary Vein Isolation - A Prospective Observational Study (AAHI Study)
Brief Title: Impact of Atrial Fibrillation Ablation on Sleep Parameters.
Acronym: AAHI
Status: Recruiting | Type: Observational
Sponsor: Primula Clinics (Other)
Responsible Party: Sponsor
Other Study IDs: KB/1641/25
Record Dates: First submitted 2025-11-13; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); OSA - Obstructive Sleep Apnea; Pulmonary Vein Isolation
Keywords: atrial fibrillation; sleep apnea; sleep apnoea; ablation; pulmonary vein isolation; pvi; snoring; choking; somnolence
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Snoring; Airway Obstruction; Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Afib scheduled for PVI, at least one risk factor for obstructive sleep apnea.

SUMMARY:
Assessment of Sleep Parameters Using Polygraphy in Patients with Paroxysmal Atrial Fibrillation Qualified for Pulmonary Vein Isolation - A Prospective Observational Study: Afib Ablation and Hypopnea Index - The "AAHI" Study

Principal Investigator:

Dr. Paweł Basiukiewicz, MD, PhD

Study Sponsor:

Primula Clinics sp. z o.o. Żyrardowska 31, 05-825 Grodzisk Mazowiecki, Poland NIP (Tax ID): 529 183 03 11

Dear Sir/Madam,

You have been invited to participate in a scientific study aimed at assessing sleep parameters in patients with atrial fibrillation undergoing rhythm-control therapy. Please read this document carefully before deciding whether to take part in the study. If you have any questions, please contact the principal investigator.

Study Objective:

To assess sleep parameters using polygraphy in the course of treatment of patients with paroxysmal atrial fibrillation qualified for pulmonary vein isolation.

Study Procedures:

The study involves four polygraphic sleep studies (two before and two after atrial fibrillation ablation), each conducted at least 7 days apart.

The polygraphic studies will record the following parameters: pulse oximetry, heart rate, respiratory movements of the chest, and airflow through the anterior nares.

The study includes only patients undergoing atrial fibrillation ablation for the first time.

Risks and Benefits:

The study is non-invasive and does not involve any direct health risks. Participation will not affect your treatment process, but it may provide valuable information about your health status.

Voluntary Participation:

Participation in the study is entirely voluntary. You may withdraw from the study at any time without providing a reason and without any impact on your ongoing medical treatment.

Personal Data Protection (GDPR):

In accordance with Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 (General Data Protection Regulation - GDPR):

The data controller is Primula Clinics sp. z o.o.

Personal data will be processed solely for the purpose of conducting this study.

Data will be stored no longer than required by law or necessary for the research purposes.

You have the right to access your data, request its correction, deletion, restriction of processing, and to object to data processing.

All data will be protected against unauthorized access.

DETAILED DESCRIPTION:
Study Title

Assessment of Sleep Parameters Using Polygraphy in Patients With Paroxysmal Atrial Fibrillation Qualified for Pulmonary Vein Isolation - A Prospective Observational Study: AFib Ablation and Hypopnea Index - The "AAHI" Study

Principal Investigator: Dr. Paweł Basiukiewicz, MD, PhD Study Sponsor: Primula Clinics sp. z o.o. Żyrardowska 31, 05-825 Grodzisk Mazowiecki, Poland NIP (Tax ID): 529 183 03 11

2. Introduction and Study Rationale

Atrial fibrillation (AFib) is the most common cardiac arrhythmia and is associated with an increased risk of cardiovascular complications and reduced quality of life. Obstructive sleep apnea (OSA) frequently coexists with AFib and may influence both the course of the arrhythmia and the effectiveness of its treatment, including catheter ablation. It is known that atrial fibrillation may exacerbate obstructive sleep apnea through mechanisms such as the loss of atrioventricular synchrony, absence of the so-called "atrial kick," tachycardia, and fluid redistribution within the body during AFib episodes.

The aim of this study is to assess changes in sleep parameters, measured by polygraphy, during the treatment course of patients with atrial fibrillation who are qualified for pulmonary vein isolation.

3. Study Objective

To assess sleep parameters using polygraphy during the course of treatment of patients with paroxysmal atrial fibrillation qualified for pulmonary vein isolation.

4. Research Hypothesis

Sleep parameters assessed via polygraphy, particularly the Apnea-Hypopnea Index (AHI), change following rhythm-control therapy.

5. Study Population

Inclusion Criteria:

Patients with atrial fibrillation who have been previously qualified for AFib ablation.

Presence of at least one risk factor for sleep apnea from the following list: diabetes, hypertension, male sex, BMI > 25, neck circumference > 42 cm in women and > 45 cm in men, upper airway obstruction, history of snoring, daytime sleepiness or fatigue, or witnessed apneic events or choking episodes during sleep.

Exclusion Criteria:

Absence of sleep apnea risk factors.

Lack of consent to participate in the study.

Study Notes:

Polygraphic assessments will be performed as a standard procedure recommended in clinical guidelines, ensuring that the study does not interfere with routine patient care.

Therefore, the study maintains an observational, non-interventional character.

6. Study Procedures

1. Before the planned AFib ablation:

   Two polygraphic studies will be performed at least 7 days apart.

   Recorded channels: pulse oximetry, heart rate, respiratory movements of the chest and abdomen using respiratory inductance plethysmography (RIP) belts, and nasal airflow (pressure) through the anterior nares.
2. After AFib ablation:

   Two polygraphic studies will be performed, at least 7 days apart, beginning one month after the ablation procedure.

   The same recording channels as above will be used.
3. Routine recommendations:

   All standard-of-care procedures, including lifestyle modification advice and non-pharmacological interventions (e.g., initiation of CPAP therapy, if indicated), will be provided to each patient in accordance with routine clinical practice.
4. Ablation procedure:

The ablation is not part of the study. It is a pre-planned, routine clinical procedure scheduled prior to study screening.

7. Methodology

Polygraphic Studies:

Certified sleep-monitoring equipment will be used (Nox polygraph, Nox Medical).

Analysis will include AHI, oxygen saturation, heart rate, and respiratory pattern assessment.

Planned Study Population: Approximately 100 participants.

Study Duration: Recruitment period estimated at 6-12 months, with the possibility of extension and inclusion of additional centers if the necessary criteria are met.

Statistical Analysis:

Comparison of pre- and post-ablation sleep parameters using appropriate statistical tests (e.g., paired t-test for parametric data or Wilcoxon test for non-parametric data).

Endpoints: Statistically significant changes in sleep parameters (particularly AHI) recorded by polygraphy.

8. Ethics

The study is observational and does not interfere with standard patient treatment.

All participants will provide written informed consent after being informed about the purpose, course, and potential benefits of the study.

The study will be conducted in accordance with the Declaration of Helsinki and approved by the local bioethics committee.

9. Results and Application

The study results may provide insight into the potential effects of rhythm-control therapy on sleep parameters in patients with atrial fibrillation. This could contribute to a better understanding of the relationship between these two conditions and to optimizing patient management.

ELIGIBILITY:
Inclusion Criteria (all must be met):

* Diagnosis of atrial fibrillation (AFib) and scheduled catheter ablation.
* Presence of at least one OSA risk factor: hypertension, male sex, BMI > 25, diabetes, excessive daytime sleepiness, snoring.

Exclusion Criteria:

- Absence of predefined sleep apnea risk factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AFib scheduled for pulmonary vein isolation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from the baseline in post ablation apnea-hypopnea index (AHI) | From baseline through study completion, an average of 1 year
  Change in apnea - hypopnea index after atrial fibrillation ablation (pulmonary vein isolation). Improvement will be assessed as a decrease in the Apnea-Hypopnea Index.
apnea - hypopnea index (AHI) change | From baseline through study completion, an average of 1 year
  Assessment of change of AHI post PVI procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Paweł S Basiukiewicz, MD, PhD, Principal Investigator — Primula Clinics
Locations (1):
- Primula Clinics, Grodzisk Mazowiecki, Poland

IPD SHARING:
Plan to Share IPD: Yes
Database with participants (DOB, HSAT data, PVI date and echocardiograhy findings)
Supporting Information: Study Protocol
Time Frame: 01.01.2026 till 01.01.2027
Access Criteria: Investigators with granted permission from PI

REFERENCES:
- [Background] Shantha G, Pelosi F, Morady F. Relationship Between Obstructive Sleep Apnoea and AF. Arrhythm Electrophysiol Rev. 2019 Jul;8(3):180-183. doi: 10.15420/aer.2019.35.2. PMID 31463055
- [Background] Linz D, Baumert M, Desteghe L, Kadhim K, Vernooy K, Kalman JM, Dobrev D, Arzt M, Sastry M, Crijns HJGM, Schotten U, Cowie MR, McEvoy RD, Heidbuchel H, Hendriks J, Sanders P, Lau DH. Nightly sleep apnea severity in patients with atrial fibrillation: Potential applications of long-term sleep apnea monitoring. Int J Cardiol Heart Vasc. 2019 Oct 18;24:100424. doi: 10.1016/j.ijcha.2019.100424. eCollection 2019 Sep. PMID 31763438
- [Background] Van Gelder IC, Rienstra M, Bunting KV, Casado-Arroyo R, Caso V, Crijns HJGM, De Potter TJR, Dwight J, Guasti L, Hanke T, Jaarsma T, Lettino M, Lochen ML, Lumbers RT, Maesen B, Molgaard I, Rosano GMC, Sanders P, Schnabel RB, Suwalski P, Svennberg E, Tamargo J, Tica O, Traykov V, Tzeis S, Kotecha D; ESC Scientific Document Group. 2024 ESC Guidelines for the management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2024 Sep 29;45(36):3314-3414. doi: 10.1093/eurheartj/ehae176. No abstract available. PMID 39210723